CLINICAL TRIAL: NCT02877979
Title: A Double-blind, Randomised, Placebo-controlled, Dose Escalation Trial to Evaluate the Safety and to Assess Local and Systemic Pharmacokinetics of DS003 Vaginal Tablets Administered to Healthy HIV-negative Women
Brief Title: Evaluate the Safety & Assess Local and Systemic PK of DS003 Vaginal Tablets Administered to Healthy HIV-negative Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: IPM 042
Record Dates: First submitted 2016-07-25; First posted 2016-08-25 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: HIV

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DS003 vaginal tablet (Experimental): participants will be randomised in a 3:1 ratio to receive either DS003 or placebo on Day 0 and Day 17.
  Interventions: Drug: DS003 vaginal tablet
- placebo (Placebo Comparator): participants will be randomised in a 3:1 ratio to receive either DS003 or placebo on Day 0 and Day 17.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DS003 vaginal tablet — The trial will be conducted in three cohorts of 12 women each. In each cohort, participants will be randomised in a 3:1 ratio to receive either DS003 or placebo on Day 0 and Day 17. In each cohort, therefore, 9 participants will receive DS003 vaginal tablets and 3 participants will receive placebo vaginal tablets.
  Arms: DS003 vaginal tablet
Drug: Placebo
  Arms: placebo

SUMMARY:
A double-blind, randomised, placebo-controlled, dose escalation trial to evaluate the safety and to assess local and systemic pharmacokinetics of ds003 vaginal tablets administered to healthy HIV-negative women.

ELIGIBILITY:
Inclusion Criteria:

Women must meet all of the following criteria to be eligible for enrolment:

1. Women ≥ 18 and ≤ 45 years of age who can give written informed consent
2. BMI of ≥ 18 and < 30 kg/m2
3. Vital signs within normal limits and no clinically significant ECG findings
4. Available for all visits and consent to follow all procedures scheduled for the trial
5. Healthy, based on medical history, vital signs, physical examination, urinalysis (dipstick and microscopy), laboratory evaluations for genital infections (bacterial vaginosis, gonorrhoea, chlamydia and trichomonas) and laboratory evaluations for haematology and biochemistry
6. HIV-negative as determined by an HIV test at the time of screening
7. On a stable form of contraception, defined as:

   * A stable oral contraceptive regimen for at least 2 months prior to enrolment, OR
   * Transdermal contraceptive patch for at least 3 months prior to enrolment, OR
   * Subcutaneous implant inserted at least 3 months prior to enrolment, OR
   * Long-acting progestins for at least 2 consecutive injections, OR An IUD inserted (with no vaginal or gynaecological complaints associated with its use) at least 3 months prior to enrolment, OR
   * Have undergone surgical sterilisation at least 3 months prior to enrolment AND be willing to use oral contraceptives if necessary to delay menstruation while taking part in the trial
8. Upon pelvic examination and colposcopy at screening and visual inspection of the cervix at the time of enrolment, the cervix and vagina appear normal as determined by the Investigator
9. Asymptomatic for urogenital infections at the time of screening (if a woman is diagnosed with any curable STI, either clinically or by laboratory test at the time of screening, she must complete the full course of treatment and have a healthy genital tract before being considered for potential re-screening)
10. Willing to refrain from the use of topical vaginal medications, vaginal products or objects, including tampons, female condoms, cotton wool, rags, diaphragms, cervical caps (or any other vaginal barrier method), douches, lubricants, vibrators/dildos, and drying agents for 7 days prior to enrolment and for the duration of the trial
11. Documentation of no abnormality on cervical cytology, including grossly bloody smear, within 90 days prior to screening
12. Willing to refrain from participation in any other research trial for the duration of this trial
13. Willing to provide adequate locator information for trial retention purposes and be reachable per local standard procedures, e.g. by home visit or telephone, or via family or close neighbour contacts (confidentiality to be maintained)
14. Willing to agree to abstain from all the following for a total of 2 days (48 hours) prior to each trial visit, and for a total of 3 days (72 hours) after the biopsy procedure:

    Penile-vaginal intercourse

    • Oral contact with her genitalia
15. Hepatitis B and C negative at the time of screening

Exclusion Criteria:

Women who meet any of the exclusion criteria below are not eligible:

1. Currently pregnant or had their last pregnancy outcome within 3 months prior to screening
2. Currently breast-feeding
3. Currently or within 2 months of participation in any other clinical research trial involving investigational or marketed products prior to screening
4. Untreated symptomatic urogenital infections, e.g. urinary tract or other sexually transmitted infections, or other gynaecological conditions such as vaginal itching, pain, or discharge, prior to enrolment
5. Have a Grade 2 or higher pelvic examination finding, according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events; Addendum 1 Female Genital Grading Table for Use in Microbicide Studies
6. History of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding, urethral obstruction, incontinence or urge incontinence
7. Current vulvar or vaginal symptoms/abnormalities that could influence the trial results
8. Cervical cytology at screening that requires cryotherapy, biopsy, treatment, or further evaluation
9. Symptomatic genital herpes simplex virus (HSV) infection or a history of genital herpetic infection
10. Any Grade 2, 3 or 4 haematology, biochemistry or urinalysis laboratory abnormality at baseline (screening) according to the current version of the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events
11. Unexplained, abnormal bleeding per vagina during or following vaginal intercourse, or gynaecologic surgery within 90 days prior to enrolment
12. Any history of anaphylaxis or severe allergy resulting in angioedema; or a history of sensitivity/allergy to latex
13. Any serious acute, chronic or progressive disease (e.g. any known history of neoplasm, cancer, diabetes, epilepsy, cardiac disease, autoimmune disease, HIV, AIDS, or blood dyscrasias), or signs of cardiac disease, renal failure, or severe malnutrition
14. Have undergone a hysterectomy
15. History of drug or substance abuse within 1 year of enrolment
16. Use of tobacco within 6 months of enrolment
17. Not willing to abstain from alcohol from 14 days prior to enrolment until completion of trial participation
18. Have had significant blood loss, or have donated or received one or more units of blood within 6 weeks prior to enrolment
19. Have a positive urine drug or positive breath alcohol screen at screening or enrolment
20. Any disease or condition (medical or surgical) that might compromise haematological, cardiovascular, pulmonary, renal, gastrointestinal, or central nervous system function; or any other conditions that might interfere with the absorption, distribution, metabolism, or excretion of the investigational product, or that would place the participant at increased risk, as determined by the Investigator
21. Regular use of, or have received, any concomitant prescription, over-the-counter, or herbal medications or nutritional supplements within 14 days prior to enrolment
22. Any condition(s) that, in the opinion of the Investigator, might interfere with adherence to trial requirements or evaluation of the trial objectives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2016-08-26 (Actual); Study Completion 2016-08-26 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of three escalating doses of DS003 (1 mg, 3 mg and 10 mg), administered in a vaginal tablet formulation, to healthy, HIV-negative female volunteers. | 12 weeks
  Gynaecological assessments, including pelvic examination and colposcopy

SECONDARY OUTCOMES:
To assess the local (vaginal fluids) and systemic (plasma) DS003 PK profile and the 24 hour cervical tissue concentration when administered in three escalating doses of a vaginal tablet formulation. | 12 weeks
  Measurement of DS003 concentrations in plasma, vaginal fluids and cervical tissue collected at various time points after administration of the vaginal tablet(s).

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Herrera C, Harman S, Aldon Y, Rogers P, Armanasco N, Ziprin P, Stieh D, Nuttall J, Shattock RJ. The entry inhibitor DS003 (BMS-599793): a BMS-806 analogue, provides superior activity as a pre-exposure prophylaxis candidate. AIDS. 2021 Oct 1;35(12):1907-1917. doi: 10.1097/QAD.0000000000002974. PMID 34101626